CLINICAL TRIAL: NCT01104805
Title: NIDA-CTN-0044: Web-delivery of Evidence-Based, Psychosocial Treatment for Substance Use Disorders Using the Therapeutic Education System (TES)
Brief Title: Web-delivery of Evidence-based, Psychosocial Treatment for Substance Use Disorders
Acronym: CTN-0044
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYSPI #6051; U10DA013035 (NIH); NIDA-CTN-0044 (Other: NIDA CTN Protocol Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Substance Abuse
Keywords: Drug Abuse; Substance Abuse; Substance Use Disorder; Addiction; Behavioral Treatment
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — TES; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Education System (TES) (Experimental): Participants randomized to this arm will replace approximately 2 hours of Standard Treatment with the Therapeutic Education System (TES) (comprised of a web-based version of the Community Reinforcement Approach and contingency management).
  Interventions: Behavioral: Therapeutic Education System (TES)
- Treatment-as-Usual (TAU) (Other): Participants randomized to TAU will receive standard treatment offered and prescribed, as usual, in the outpatient substance abuse treatment program.
  Interventions: Behavioral: Treatment-as-Usual (TAU)

INTERVENTIONS:
Behavioral: Therapeutic Education System (TES) — Participants will received modified treatment-as-usual plus the computerized psychosocial intervention (Therapeutic Education System), including contingency management. Participants will be asked to use the self-directed TES intervention twice weekly and will be asked to complete 2 modules during each session (for a total of 4 modules per week) during the 12-week intervention. Participants will receive incentives contingent primarily upon abstinence from drugs of abuse and, secondarily, upon completion of TES modules.
  Other Names: Therapeutic Education System; TES
  Arms: Therapeutic Education System (TES)
Behavioral: Treatment-as-Usual (TAU) — Participants in this condition will receive TAU, consisting of standard treatment offered at each collaborating CTP and will reflect the model of treatment typically provided to most individuals in outpatient, community-based substance abuse treatment settings in the U.S. These sessions will consist of a combination of group and individual counseling.
  Other Names: Treatment as Usual; TAU; Standard Treatment
  Arms: Treatment-as-Usual (TAU)

SUMMARY:
The main objective of this study is to evaluate the effectiveness of including an interactive, web-based version of the Community Reinforcement Approach (CRA), called the Therapeutic Education System (TES), as part of community-based, outpatient substance abuse treatment.

DETAILED DESCRIPTION:
The principal objective of the planned trial is to evaluate the effectiveness of including an interactive, web-based version of the Community Reinforcement Approach (CRA), called the Therapeutic Education System (TES), as part of community-based, outpatient substance abuse treatment. CRA is a cognitive-behavioral intervention which seeks to give patients skills to achieve and maintain abstinence and improve social functioning and is often paired with contingency management, where patients earn rewards contingent upon drug negative urines. CRA is an intensive treatment, generally delivered in individual sessions 2 to 3 times per week. Thus, it is expensive and time-consuming to deliver, to train clinical staff, and to provide supervision to maintain clinical staff skill. However, because CRA is oriented toward knowledge and skills, it lends itself to being delivered by computer, using computer-interactive learning technologies.

Individuals accepted into community-based outpatient treatment for substance use disorders (excluding those receiving opioid pharmacotherapy for opioid dependence) will be eligible to participate. This is a multi-site, controlled trial, using NIDA's Clinical Trials Network platform, at approximately 10 Community Treatment Programs, in which participants (N = approximately 500) will be randomized to receive 12 weeks of either: (1) Treatment-as-Usual (TAU), reflecting standard treatment at the collaborating treatment programs in which participants are enrolled, or (2) a modification of TAU which includes access to the TES. It is hypothesized that access to TES will improve substance use outcome and retention in outpatient treatment.

Computer interactive interventions like TES have the potential to deliver science-based psychosocial treatments with high fidelity and cost-effectiveness while conserving clinician time to focus on monitoring and addressing patients' needs. If found to be effective, TES could substantially advance the substance abuse treatment system by improving quality of care delivered, increasing availability of treatment slots by extending and leveraging the efforts of clinical staff, and projecting treatment to rural and other underserved areas.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18 years or older, accepted for outpatient, substance abuse treatment at a participating study site.
* Self-report any substance use problem (including alcohol, as long as they also report other drug use in addition to alcohol).
* Self-report recent drug use.
* Within 30 days of initiating treatment at a collaborating study site.
* Self-report a planned substance abuse treatment episode of at least 3 months.

Exclusion Criteria:

* Receiving opioid replacement medication.
* Plan to move out of the area within the next 3 months.
* Insufficient ability to provide informed consent.
* Insufficient ability to use English to participate meaningfully in the consent process, the interventions or research assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduced Substance Use and Improved Treatment Retention | 12-week Treatment Phase
  Compared to patients assigned to Treatment as Usual (TAU), patients assigned to modified TAU plus the Therapeutic Education System (Modified TAU + TES) will have:
  1. reduced substance use (measured by a combination of self-report confirmed by urine toxicology) and
  2. better retention in treatment at their community-based treatment programs.

SECONDARY OUTCOMES:
Effectiveness | 12-week treatment phase, 3- and 6-months post treatment
  To evaluate the relative effectiveness of TAU vs. modified TAU + TES on several secondary outcome measures, including measures of HIV risk behavior, psychosocial functioning (in areas of criminal activity, health status improvement, psychological status, family/social relationships, and employment, and treatment acceptability (based on participant feedback).
Sustained outcome | 3- and 6-months post treatment
  To evaluate if improved substance use and retention outcomes are maintained 3- and 6-months post-intervention.
Economic Analysis | 12-week treatment phase, 3- and 6-months post treatment
  To perform a comprehensive economic analysis of including TES in TAU to inform decisions regarding adoption of this new therapeutic tool (assessing incremental costs per increased abstinence time and quality adjusted life year). The economic analyses are clinically important, as even if the computerized intervention is shown to be effective, it may not be adopted in community-based treatment programs unless it is shown to be cost-effective due to the considerable financial constraints in such treatment settings.
Coping Skills | 12-week treatment phase, 3- and 6-months post treatment
  To examine coping skills acquisition as a treatment process factor that may underlie changes observed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Nunes, MD, Principal Investigator — NIDA Clinical Trials Network - Long Island Regional Node
Locations (10):
- United States (10):
  - MCCA: Midwestern CT Council on Alcoholism, Danbury, Connecticut
  - The Center for Drug Free Living, Orlando, Florida
  - Hina Mauka, Waipahu, Hawaii
  - Midtown Community Mental Health Center, Indianapolis, Indiana
  - HARBEL Prevention and Recovery Center, Baltimore, Maryland
  - Stanley Street Treatment and Resources (SSTAR), Fall River, Massachusetts
  - Project Outreach, West Hempstead, New York
  - Willamette Family, Inc., Eugene, Oregon
  - Homeward Bound, Dallas, Texas
  - Evergreen Manor, Everett, Washington

REFERENCES:
- [Derived] Luderer HF, Campbell ANC, Nunes EV, Enman NM, Xiong X, Gerwien R, Maricich YA. Engagement patterns with a digital therapeutic for substance use disorders: Correlations with abstinence outcomes. J Subst Abuse Treat. 2022 Jan;132:108585. doi: 10.1016/j.jsat.2021.108585. Epub 2021 Jul 30. PMID 34366201
- [Derived] Murphy SM, Campbell AN, Ghitza UE, Kyle TL, Bailey GL, Nunes EV, Polsky D. Cost-effectiveness of an internet-delivered treatment for substance abuse: Data from a multisite randomized controlled trial. Drug Alcohol Depend. 2016 Apr 1;161:119-26. doi: 10.1016/j.drugalcdep.2016.01.021. Epub 2016 Jan 30. PMID 26880594
- [Derived] Cochran G, Stitzer M, Campbell AN, Hu MC, Vandrey R, Nunes EV. Web-based treatment for substance use disorders: differential effects by primary substance. Addict Behav. 2015 Jun;45:191-4. doi: 10.1016/j.addbeh.2015.02.002. Epub 2015 Feb 8. PMID 25697725
- [Derived] Mitchell SG, Schwartz RP, Alvanzo AA, Weisman MS, Kyle TL, Turrigiano EM, Gibson ML, Perez L, McClure EA, Clingerman S, Froias A, Shandera DR, Walker R, Babcock DL, Bailey GL, Miele GM, Kunkel LE, Norton M, Stitzer ML. The Use of Technology in Participant Tracking and Study Retention: Lessons Learned From a Clinical Trials Network Study. Subst Abus. 2015;36(4):420-6. doi: 10.1080/08897077.2014.992565. Epub 2015 Feb 11. PMID 25671593
- [Derived] Cochran G, Stitzer M, Nunes EV, Hu MC, Campbell A. Clinically relevant characteristics associated with early treatment drug use versus abstinence. Addict Sci Clin Pract. 2014 Apr 4;9(1):6. doi: 10.1186/1940-0640-9-6. PMID 24708748
- See also: National Institute on Drug Abuse, Clinical Trials Network — http://www.drugabuse.gov/CTN/